CLINICAL TRIAL: NCT06509698
Title: Comparative Effects of Virtual Reality and Frenkel's Exercises on Balance, Gait and Quality of Life in Patients With Stroke.
Brief Title: Comparative Effects of Virtual Reality and Frenkel's Exercises in Patients With Stroke.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0284 Aqsa
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Balance; Berg balance scale; Frenkel's exercises; gait; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): Virtual reality used for balance, gait and quality of life the treatment will be given with the frequency of 3 times per week for 6 weeks. Warmup period, Instruct the patient/participants, Gaming time (20 minutes), cool down period (5 minutes).
  Treatment sessions will be of 30 minutes with short resting intervals.
  Interventions: Other: virtual reality
- Frenkel's exercise (Active Comparator): Frenkel's exercise used for balance, gait and quality of life Frenkel's exercise, the treatment will be given with the frequency of 3 times per week for 6 weeks.
  Warmup period (5 minutes), frenkel's exercise (20 minutes), cool down period (5 minutes).
  Treatment sessions will be of 30 minutes with short resting intervals.
  Interventions: Other: Frenkel's exercise

INTERVENTIONS:
Other: virtual reality — STEP I: For the warm-up, the examiner will perform passive stretching exercises to maintain the range of motion. STEP II: The patient will receive the game instructions by the examiner. STEP III: The patient will play the Adventure games and Sport games including tennis, boxing and kicking. virtual reality (20 minutes) using Nintendo Wii®, Wii Fit game will be used to stimulate and reinforce the improvement of balance and gait and enhance the quality of life.(30) Balance game: Soccer Heading, Penguin Slides, Balance Bubble, Torso Twists, and Single Leg Stance. Motor function: Boxing, Kicking, Tennis and Bowling Aerobic Games: 2-P run, advanced step, Title city and Basic Run. Step IV: (cool-down): Same as step one.
  Arms: virtual reality
Other: Frenkel's exercise — Frenkel's activities, which included learning how to turn around, sit down, and get up using a variety of commonplace objects like chairs, beds, or traces drawn on the floor, as well as learning how to walk with upper limb coordination. This is a typical workout regimen used in testing and rehabilitation centers. Patients engaged in the following activities, each activity time is 1.5 minutes
  Arms: Frenkel's exercise

SUMMARY:
To compare the effects of Virtual reality and Frenkel's exercises on balance, gait and quality of life in patients with stroke.

DETAILED DESCRIPTION:
This randomized Control trial will be conducted at Islam central hospital, Sialkot over a duration of 7 months after approval of synopsis. 36 Participants who meet the inclusion criteria will be further divided into 2 groups. The treatment will be given with the frequency of 3 times per week for 6 weeks. Treatment sessions will be of 30 minutes with short resting intervals. Data will be collected using various assessment tools including, berg balance scale, time-up and stroke-specific quality of life. Pre-intervention assessment will be conducted before starting the treatment protocol and post assessment after 6 weeks of treatment. The data will be analyzed using SPSS version 28 for Windows software. Statistical significance will be set at p = 0.05. Normality of data will be assessed through Kolmogorov Smirnov test. Difference between pre-treatment and post-treatment readings will be calculated using Paired sample t-test for parametric data. For non-parametric data Wilcoxon test will be used. Independent sample t-test will be used for parametric data and Mann Whitney test will be used for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

1- Age 40-65 years. 2. Stroke patients with both genders. 3. Subacute stroke patients will be included. 4. Survivors of ischemic stroke. 5. No prior experience with VR-based rehabilitation. 6. Patients with ≥24 Mini-Mental State Exam score.

Exclusion Criteria:

1. Patient with serious behavioral problems or mental health.
2. Patients with recent lower extremity deep vein thrombosis, quadriplegia, Parkinson's disease, lower limb fractures, or recent myocardial infarction.
3. Patients with malignant tumor, or other unstable condition.
4. Participants with ENT defect, hearing, majorly affected vision(blindness), cataract, glaucoma, loss of vision.
5. Subjects with diagnosed vestibular disease.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
berg balance scale | 6-weeks
  The BBS is an instrument that assesses functional balance performance in older adults using 14 tasks: sitting to standing, standing unsupported, sitting unsupported, standing to sitting, transfers, standing with eyes closed, standing with feet together, reaching forward with outstretched arm, retrieving object from floor, turning to look behind, turning 360 degrees, placing the foot alternately on a step, standing with 1 foot in front, and standing on 1 foot.18 The maximum score is 56 points, representing normal balance. Each item is scored from 0 (unable to perform) to 4 (normal performance)
time up and go | 6-weeks
  A straightforward performance test called the Timed-Up-and-Go (TUG) is frequently used to evaluate stroke patients' functional mobility and may be able to reveal some information on turning movement. The patient was really instructed to get up from a seated posture, walk three metres, turn around 180 degrees, walk three metres back, turn around 180 degrees, and then sit down once again. It is a viable tool to monitor walkable stroke patients because it is an easy-to-administer, quick test with good intra- and inter-rater reliability, strong convergent validity, and sensitivity to modest changes.4. The amount of time the patient needs to do the task in total determines their score. In fact, the TUG integrates several mobility functions, and its various subcomponents include intricate tasks.
stroke specific quality of life | 6-weeks
  A disease-specific patient-reported outcome measure called the SSQOL was created to evaluate the quality of life for stroke survivors. The 48 items are categorized into 12 domains: job, language, mobility, thinking, personality, mood, family roles, social roles, energy, self-care, vision, and upper extremity function. Each domain has three to six items. Likert scale answers are used for the items, with the least impacted item receiving a score of one and the unaffected item receiving a score of five. The questionnaire has a maximum total score of 245 and a minimum score of 49. A quality of life score of 60% of the maximum value indicates poor life.

CONTACTS AND LOCATIONS:
Overall Officials: Alveena Fatima, Ms.NMPT, Principal Investigator — Riphah International University
Locations (1):
- Alveena fatima, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng X, Wu X, Liu Z, Wang J, Wang K, Yin J, Wang X. The Influences of Tai Chi on Balance Function and Exercise Capacity among Stroke Patients: A Meta-Analysis. Evid Based Complement Alternat Med. 2021 Feb 24;2021:6636847. doi: 10.1155/2021/6636847. eCollection 2021. PMID 33708256
- [Background] Beckwee D, Lefeber N, Bautmans I, Cuypers L, De Keersmaecker E, De Raedt S, Kerckhofs E, Nagels G, Njemini R, Perkisas S, Scheys E, Swinnen E. Muscle changes after stroke and their impact on recovery: time for a paradigm shift? Review and commentary. Top Stroke Rehabil. 2021 Mar;28(2):104-111. doi: 10.1080/10749357.2020.1783916. Epub 2020 Jun 26. PMID 32588773
- [Background] Duan J, Gao S, Tu S, Lenahan C, Shao A, Sheng J. Pathophysiology and Therapeutic Potential of NADPH Oxidases in Ischemic Stroke-Induced Oxidative Stress. Oxid Med Cell Longev. 2021 Mar 9;2021:6631805. doi: 10.1155/2021/6631805. eCollection 2021. PMID 33777315
- [Background] Hsu CC, Fu TC, Huang SC, Chen CP, Wang JS. Increased serum brain-derived neurotrophic factor with high-intensity interval training in stroke patients: A randomized controlled trial. Ann Phys Rehabil Med. 2021 Jul;64(4):101385. doi: 10.1016/j.rehab.2020.03.010. Epub 2020 May 11. PMID 32344098
- [Background] Feske SK. Ischemic Stroke. Am J Med. 2021 Dec;134(12):1457-1464. doi: 10.1016/j.amjmed.2021.07.027. Epub 2021 Aug 27. PMID 34454905
- [Background] Uwishema O, Berjaoui C, Correia IFS, Anis H, Karabulut E, Essayli D, Mhanna M, Oluyemisi A. Current management of acute ischemic stroke in Africa: A review of the literature. Eur J Neurol. 2022 Nov;29(11):3460-3465. doi: 10.1111/ene.15495. Epub 2022 Jul 26. PMID 35837810
- [Background] Ullah I, Arsh A, Zahir A, Jan S. Motor relearning program along with electrical stimulation for improving upper limb function in stroke patients: A quasi experimental study. Pak J Med Sci. 2020 Nov-Dec;36(7):1613-1617. doi: 10.12669/pjms.36.7.2351. PMID 33235584
- [Background] Lau LH, Lew J, Borschmann K, Thijs V, Ekinci EI. Prevalence of diabetes and its effects on stroke outcomes: A meta-analysis and literature review. J Diabetes Investig. 2019 May;10(3):780-792. doi: 10.1111/jdi.12932. Epub 2018 Oct 13. PMID 30220102
- [Background] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236